CLINICAL TRIAL: NCT03040882
Title: Effectiveness of Cotton Sock in Pediatric Patients With Leg-foot Splint After Surgery for Correction of the Foot, in Reducing the Incidence of Cutaneous Lesions. Randomized Controlled Trial.
Brief Title: Cotton Sock in Pediatric Patients With Leg-foot Splint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0014868
Record Dates: First submitted 2017-02-01; First posted 2017-02-02 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2017-01

CONDITIONS: Flat Foot
MeSH Terms: conditions — Flatfoot | interventions — Compression Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cotton sock (Experimental)
  Interventions: Other: cotton sock
- Elastic Compression Wraps (Active Comparator)
  Interventions: Other: Elastic Compression Wraps

INTERVENTIONS:
Other: cotton sock — Application of a cotton sock in the immediate postoperative period before applied the Walker
  Arms: cotton sock
Other: Elastic Compression Wraps — Application of an Elastic Compression Wraps in the lower limb in the immediate postoperative period before applied the Walker (standard care)
  Arms: Elastic Compression Wraps

SUMMARY:
The post-operative treatment of pediatric patients operated for the correction of flat foot, sees today the use of preformed leg-foot splint (Walker) as an alternative to the application of plaster casts. The change of the immobilization system has led to the appearance of problems of tolerability in particular in the skin. The problems persist also after placing a polyurethane foam dress at the heel in the immediate postoperative period. The aim of this study is to evaluate the effectiveness of a cotton sock applied inside the leg-foot splint in children operated vs the Elastic Compression Wraps in reducing the incidence of cutaneous lesions.

ELIGIBILITY:
Inclusion Criteria:

* Children aged > 3 years
* Treated for flat foot
* Children with intact skin at the heel

Exclusion Criteria:

* Caregivers who cannot speak Italian
* Those who refuse to give their consent to take part in the study
* Patients with lower limb casts

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Heel Pressure Sores | every day until discharge (expected average of 3 days).
  • Numbers of Participants With Heel Pressure Sores of all grade Detected According to the Classification of the Scale of the National Pressure Ulcer Advisory Panel -N.P.U.A.P.

SECONDARY OUTCOMES:
Pain | up to the first 3 days post intervention
  Pain Score on the "Numeric Rating Scale"

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Guerra, RN, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No